CLINICAL TRIAL: NCT01603407
Title: Duchenne Muscular Dystrophy: Double-blind Randomized Trial to Find Optimum Steroid Regimen
Brief Title: Finding the Optimum Regimen for Duchenne Muscular Dystrophy
Acronym: FOR-DMD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Newcastle University (Other); University Medical Center Freiburg (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Robert Griggs, MD, Professor of Neurology, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: U01NS061799 (NIH); 2010-023744-33 (EudraCT Number); U01NS061799 (NIH); 46102316 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2012-04-03; First posted 2012-05-23 (Estimated); Results first posted 2022-08-12 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: prednisone; deflazacort; muscular dystrophy; neuromuscular disease; multi-center
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Muscular Dystrophies; Neuromuscular Diseases | interventions — Prednisone; deflazacort

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Daily prednisone (Experimental): daily prednisone (0.75 mg/kg/day)
  Interventions: Drug: Prednisone
- Intermittent prednisone (Experimental): intermittent prednisone (0.75 mg/kg/day, 10 days on, 10 days off)
  Interventions: Drug: Prednisone
- Daily deflazacort (Experimental): daily deflazacort (0.9 mg/kg/day
  Interventions: Drug: Deflazacort

INTERVENTIONS:
Drug: Prednisone — daily prednisone (0.75 mg/kg/day) tablets for 36-60 months
  Arms: Daily prednisone
Drug: Prednisone — intermittent prednisone (0.75 mg/kg/day, 10 days on, 10 days off) tablets for 36 to 60 months
  Arms: Intermittent prednisone
Drug: Deflazacort — daily deflazacort (0.9 mg/kg/day) tablets for 36-60 months
  Arms: Daily deflazacort

SUMMARY:
The Finding the Optimum Regimen for Duchenne Muscular Dystrophy (FOR DMD) study will compare three ways of giving corticosteroids to boys with Duchenne muscular dystrophy (DMD) to determine which of the three ways increases muscle strength the most, and which causes the fewest side effects. Using the results of this study, the investigators aim to provide patients and families with clearer information about the best way to take these drugs.

DETAILED DESCRIPTION:
Boys with Duchenne muscular dystrophy experience progressive muscle weakness as they grow up. Corticosteroids are currently the only medicine that has been shown to increase muscle strength in boys with DMD. Benefits include an increase in the length of time that boys could continue to walk, reduction in the development of curvature of the spine, a longer time of adequate breathing, and possible protection against the development of heart problems.

Doctors have tried different ways of prescribing corticosteroids in order to decrease undesirable side effects of the drug. No controlled, long-term study has ever looked at the effects of different corticosteroids to see which one improves strength the most and which one causes the fewest side effects, over a period of time. Different doctors in different countries prescribe the drugs in different ways, and some do not prescribe corticosteroids at all.

The FOR DMD study will enroll boys with DMD ages 4-7. The study will look at three ways of taking the following corticosteroids by the mouth to determine which increases muscle strength the most, and which causes the fewest side effects:

1. Prednisone 0.75mg/kg/day
2. Prednisone 0.75mg/kg/day switching between 10 days on and 10 days off treatment
3. Deflazacort 0.9mg/kg/day.

The study will take place at 40 academic medical centers in the United States, Canada, United Kingdom, Germany and Italy.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of signed and dated informed consent form.
* Confirmed diagnosis of Duchenne muscular dystrophy
* Age greater than or equal to 4 years and less than 8 years old
* Ability to rise independently from floor, from supine to standing
* Willingness and ability to comply with scheduled visits, drug administration plan and study procedures
* Ability to maintain reproducible FVC measurements.

Exclusion Criteria:

* History of major renal or hepatic impairment, immunosuppression or other contraindications to corticosteroid therapy.
* History of chronic systemic fungal or viral infections. Acute bacterial infection(including TB) would exclude from enrolment until the infection had been appropriately treated and resolved.
* Diabetes mellitus.
* Idiopathic hypercalcuria.
* Lack of chicken pox immunity and refusal to undergo immunization.
* Evidence of symptomatic cardiomyopathy at screening assessment (one to three months prior to the baseline visit). Asymptomatic cardiac abnormality on investigation would not be an exclusion.
* Current or previous treatment (greater than four consecutive weeks of oral therapy) with corticosteroids or other immunosuppressive treatments for DMD or other recurrent indications (e.g., asthma), unless approved by FOR-DMD Team (i.e., concurrent participation in another allowed DMD trial).
* Inability to take tablets, as assessed by the site investigator by the end of the screening period (the screening period ranges from one to three months prior to the baseline visit).
* Allergy/sensitivity to study drugs or their formulations including lactose and/or sucrose intolerance.
* Severe behavioral problems, including severe autism.
* Previous or ongoing medical condition, medical history, physical findings or laboratory abnormalities that could affect safety, make it unlikely that treatment and follow up will be correctly completed or impair the assessment of study results, in the judgment of the site investigator.
* Weight of less than 13 kilograms.
* Exposure to any investigational drug currently or within 3 months prior to start of study treatment.

Ages: 4 Years to 7 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 196 (Actual)
Dates: Start 2013-01; Primary Completion 2019-11 (Actual); Study Completion 2019-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert C. Griggs, MD, Principal Investigator — University of Rochester; Kate Bushby, MD, Principal Investigator — Newcastle University
Locations (32):
- United States (14):
  - University of California Los Angeles (UCLA) Medical Center, Los Angeles, California
  - University of California Davis Medical Center, Sacramento, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Nemours Children's Hospital, Orlando, Florida
  - Ann and Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Boston Children's Hospital, Boston, Massachusetts
  - University of New Mexico Health Science Center, Albuquerque, New Mexico
  - University of Rochester Medical Center, Rochester, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Nationwide Children's Hospital, Columbus, Ohio
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Vanderbilt Children's Hospital, Nashville, Tennessee
  - University of Utah Medical Center, Salt Lake City, Utah
- Canada (3):
  - Alberta Children's Hospital, Calgary, Alberta
  - Children's Hospital London Health Sciences Centre, London, Ontario
  - Children's Hospital of Eastern Ontario (CHEO), Ottawa, Ontario
- Germany (4):
  - Children's Hospital, Technical University Dresden, Dresden
  - University Hospital of Essen, Essen
  - University Medical Center Freiburg, Freiburg im Breisgau
  - Children's University Hospital, Göttingen, Göttingen
- Italy (4):
  - University of Messina AOU Policlinico Gaetano Martino, Messina
  - C. Besta Neurological Institute Foundation, Milan
  - University of Padova School of Medicine, Padua
  - Neuromuscular Center University of Turin, Torino
- United Kingdom (7):
  - The General Infirmary at Leeds, Leeds, England
  - Greater Glasgow and Clyde NHS Yorkhill Hospital, Glasgow, Scotland
  - Heart of England NHS Foundation Trust Birmingham Heartland's Hospital, Birmingham
  - Alder Hey Children's Hospital NHS Trust, Liverpool
  - Great Ormond Street Hospital for Children NHS Trust, London
  - Royal Manchester Children's Hospital, Manchester
  - Institute of Human Genetics, International Centre for Life, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Angelini C, Pegoraro E, Turella E, Intino MT, Pini A, Costa C. Deflazacort in Duchenne dystrophy: study of long-term effect. Muscle Nerve. 1994 Apr;17(4):386-91. doi: 10.1002/mus.880170405. PMID 8170484
- [Background] Atkinson MJ, Sinha A, Hass SL, Colman SS, Kumar RN, Brod M, Rowland CR. Validation of a general measure of treatment satisfaction, the Treatment Satisfaction Questionnaire for Medication (TSQM), using a national panel study of chronic disease. Health Qual Life Outcomes. 2004 Feb 26;2:12. doi: 10.1186/1477-7525-2-12. PMID 14987333
- [Background] Backman E, Henriksson KG. Low-dose prednisolone treatment in Duchenne and Becker muscular dystrophy. Neuromuscul Disord. 1995 May;5(3):233-41. doi: 10.1016/0960-8966(94)00048-e. PMID 7633189
- [Background] Bianchi ML. How to manage osteoporosis in children. Best Pract Res Clin Rheumatol. 2005 Dec;19(6):991-1005. doi: 10.1016/j.berh.2005.06.006. PMID 16301193
- [Background] Biggar WD, Bachrach LK, Henderson RC, Kalkwarf H, Plotkin H, Wong BL. Bone health in Duchenne muscular dystrophy: a workshop report from the meeting in Cincinnati, Ohio, July 8, 2004. Neuromuscul Disord. 2005 Jan;15(1):80-5. doi: 10.1016/j.nmd.2004.09.010. No abstract available. PMID 15639125
- [Background] Biggar WD, Gingras M, Fehlings DL, Harris VA, Steele CA. Deflazacort treatment of Duchenne muscular dystrophy. J Pediatr. 2001 Jan;138(1):45-50. doi: 10.1067/mpd.2001.109601. PMID 11148511
- [Background] Biggar WD, Harris VA, Eliasoph L, Alman B. Long-term benefits of deflazacort treatment for boys with Duchenne muscular dystrophy in their second decade. Neuromuscul Disord. 2006 Apr;16(4):249-55. doi: 10.1016/j.nmd.2006.01.010. Epub 2006 Mar 20. PMID 16545568
- [Background] Biggar WD, Politano L, Harris VA, Passamano L, Vajsar J, Alman B, Palladino A, Comi LI, Nigro G. Deflazacort in Duchenne muscular dystrophy: a comparison of two different protocols. Neuromuscul Disord. 2004 Sep;14(8-9):476-82. doi: 10.1016/j.nmd.2004.05.001. PMID 15336688
- [Background] Brooke MH, Fenichel GM, Griggs RC, Mendell JR, Moxley R, Miller JP, Province MA. Clinical investigation in Duchenne dystrophy: 2. Determination of the "power" of therapeutic trials based on the natural history. Muscle Nerve. 1983 Feb;6(2):91-103. doi: 10.1002/mus.880060204. PMID 6343858
- [Background] Brooke MH, Fenichel GM, Griggs RC, Mendell JR, Moxley RT 3rd, Miller JP, Kaiser KK, Florence JM, Pandya S, Signore L, et al. Clinical investigation of Duchenne muscular dystrophy. Interesting results in a trial of prednisone. Arch Neurol. 1987 Aug;44(8):812-7. doi: 10.1001/archneur.1987.00520200016010. PMID 3632393
- [Background] Brooke MH, Fenichel GM, Griggs RC, Mendell JR, Moxley R, Florence J, King WM, Pandya S, Robison J, Schierbecker J, et al. Duchenne muscular dystrophy: patterns of clinical progression and effects of supportive therapy. Neurology. 1989 Apr;39(4):475-81. doi: 10.1212/wnl.39.4.475. PMID 2927672
- [Background] Bushby K, Muntoni F, Urtizberea A, Hughes R, Griggs R. Report on the 124th ENMC International Workshop. Treatment of Duchenne muscular dystrophy; defining the gold standards of management in the use of corticosteroids. 2-4 April 2004, Naarden, The Netherlands. Neuromuscul Disord. 2004 Sep;14(8-9):526-34. doi: 10.1016/j.nmd.2004.05.006. No abstract available. PMID 15336694
- [Background] Bushby K, Muntoni F, Bourke JP. 107th ENMC international workshop: the management of cardiac involvement in muscular dystrophy and myotonic dystrophy. 7th-9th June 2002, Naarden, the Netherlands. Neuromuscul Disord. 2003 Feb;13(2):166-72. doi: 10.1016/s0960-8966(02)00213-4. No abstract available. PMID 12565916
- [Background] Bushby K, Finkel R, Birnkrant DJ, Case LE, Clemens PR, Cripe L, Kaul A, Kinnett K, McDonald C, Pandya S, Poysky J, Shapiro F, Tomezsko J, Constantin C; DMD Care Considerations Working Group. Diagnosis and management of Duchenne muscular dystrophy, part 1: diagnosis, and pharmacological and psychosocial management. Lancet Neurol. 2010 Jan;9(1):77-93. doi: 10.1016/S1474-4422(09)70271-6. Epub 2009 Nov 27. PMID 19945913
- [Background] Bushby K, Finkel R, Birnkrant DJ, Case LE, Clemens PR, Cripe L, Kaul A, Kinnett K, McDonald C, Pandya S, Poysky J, Shapiro F, Tomezsko J, Constantin C; DMD Care Considerations Working Group. Diagnosis and management of Duchenne muscular dystrophy, part 2: implementation of multidisciplinary care. Lancet Neurol. 2010 Feb;9(2):177-89. doi: 10.1016/S1474-4422(09)70272-8. Epub 2009 Nov 27. PMID 19945914
- [Background] Carter GT, McDonald CM. Preserving function in Duchenne dystrophy with long-term pulse prednisone therapy. Am J Phys Med Rehabil. 2000 Sep-Oct;79(5):455-8. doi: 10.1097/00002060-200009000-00009. PMID 10994887
- [Background] Collett BR, Ohan JL, Myers KM. Ten-year review of rating scales. V: scales assessing attention-deficit/hyperactivity disorder. J Am Acad Child Adolesc Psychiatry. 2003 Sep;42(9):1015-37. doi: 10.1097/01.CHI.0000070245.24125.B6. PMID 12960702
- [Background] Collett BR, Ohan JL, Myers KM. Ten-year review of rating scales. VI: scales assessing externalizing behaviors. J Am Acad Child Adolesc Psychiatry. 2003 Oct;42(10):1143-70. doi: 10.1097/00004583-200310000-00006. PMID 14560165
- [Background] Connolly AM, Schierbecker J, Renna R, Florence J. High dose weekly oral prednisone improves strength in boys with Duchenne muscular dystrophy. Neuromuscul Disord. 2002 Dec;12(10):917-25. doi: 10.1016/s0960-8966(02)00180-3. PMID 12467746
- [Background] Duboc D, Meune C, Lerebours G, Devaux JY, Vaksmann G, Becane HM. Effect of perindopril on the onset and progression of left ventricular dysfunction in Duchenne muscular dystrophy. J Am Coll Cardiol. 2005 Mar 15;45(6):855-7. doi: 10.1016/j.jacc.2004.09.078. PMID 15766818
- [Background] Dubowitz V, Kinali M, Main M, Mercuri E, Muntoni F. Remission of clinical signs in early duchenne muscular dystrophy on intermittent low-dosage prednisolone therapy. Eur J Paediatr Neurol. 2002;6(3):153-9. doi: 10.1053/ejpn.2002.0583. PMID 12363102
- [Background] Eagle M, Baudouin SV, Chandler C, Giddings DR, Bullock R, Bushby K. Survival in Duchenne muscular dystrophy: improvements in life expectancy since 1967 and the impact of home nocturnal ventilation. Neuromuscul Disord. 2002 Dec;12(10):926-9. doi: 10.1016/s0960-8966(02)00140-2. PMID 12467747
- [Background] Fenichel GM, Florence JM, Pestronk A, Mendell JR, Moxley RT 3rd, Griggs RC, Brooke MH, Miller JP, Robison J, King W, et al. Long-term benefit from prednisone therapy in Duchenne muscular dystrophy. Neurology. 1991 Dec;41(12):1874-7. doi: 10.1212/wnl.41.12.1874. PMID 1745340
- [Background] Fenichel GM, Mendell JR, Moxley RT 3rd, Griggs RC, Brooke MH, Miller JP, Pestronk A, Robison J, King W, Signore L, et al. A comparison of daily and alternate-day prednisone therapy in the treatment of Duchenne muscular dystrophy. Arch Neurol. 1991 Jun;48(6):575-9. doi: 10.1001/archneur.1991.00530180027012. PMID 2039377
- [Background] Follmann D. Multivariate tests for multiple endpoints in clinical trials. Stat Med. 1995 Jun 15;14(11):1163-75. doi: 10.1002/sim.4780141103. PMID 7667558
- [Background] Griggs RC, Moxley RT 3rd, Mendell JR, Fenichel GM, Brooke MH, Pestronk A, Miller JP, Cwik VA, Pandya S, Robison J, et al. Duchenne dystrophy: randomized, controlled trial of prednisone (18 months) and azathioprine (12 months). Neurology. 1993 Mar;43(3 Pt 1):520-7. doi: 10.1212/wnl.43.3_part_1.520. PMID 8450994
- [Background] Griggs RC, Moxley RT 3rd, Mendell JR, Fenichel GM, Brooke MH, Pestronk A, Miller JP. Prednisone in Duchenne dystrophy. A randomized, controlled trial defining the time course and dose response. Clinical Investigation of Duchenne Dystrophy Group. Arch Neurol. 1991 Apr;48(4):383-8. doi: 10.1001/archneur.1991.00530160047012. PMID 2012511
- [Background] Hinton VJ, Nereo NE, Fee RJ, Cyrulnik SE. Social behavior problems in boys with Duchenne muscular dystrophy. J Dev Behav Pediatr. 2006 Dec;27(6):470-6. doi: 10.1097/00004703-200612000-00003. PMID 17164619
- [Background] Hopke PK, Liu C, Rubin DB. Multiple imputation for multivariate data with missing and below-threshold measurements: time-series concentrations of pollutants in the Arctic. Biometrics. 2001 Mar;57(1):22-33. doi: 10.1111/j.0006-341x.2001.00022.x. PMID 11252602
- [Background] Kinali M, Mercuri E, Main M, Muntoni F, Dubowitz V. An effective, low-dosage, intermittent schedule of prednisolone in the long-term treatment of early cases of Duchenne dystrophy. Neuromuscul Disord. 2002 Oct;12 Suppl 1:S169-74. doi: 10.1016/s0960-8966(02)00097-4. PMID 12206813
- [Background] Lippuner K, Casez JP, Horber FF, Jaeger P. Effects of deflazacort versus prednisone on bone mass, body composition, and lipid profile: a randomized, double blind study in kidney transplant patients. J Clin Endocrinol Metab. 1998 Nov;83(11):3795-802. doi: 10.1210/jcem.83.11.5235. PMID 9814449
- [Background] Little R, Yau L. Intent-to-treat analysis for longitudinal studies with drop-outs. Biometrics. 1996 Dec;52(4):1324-33. PMID 8962456
- [Background] Loftus J, Allen R, Hesp R, David J, Reid DM, Wright DJ, Green JR, Reeve J, Ansell BM, Woo PM. Randomized, double-blind trial of deflazacort versus prednisone in juvenile chronic (or rheumatoid) arthritis: a relatively bone-sparing effect of deflazacort. Pediatrics. 1991 Sep;88(3):428-36. PMID 1881719
- [Background] Lunceford JK, Davidian M. Stratification and weighting via the propensity score in estimation of causal treatment effects: a comparative study. Stat Med. 2004 Oct 15;23(19):2937-60. doi: 10.1002/sim.1903. PMID 15351954
- [Background] Manzur AY, Kuntzer T, Pike M, Swan A. Glucocorticoid corticosteroids for Duchenne muscular dystrophy. Cochrane Database Syst Rev. 2004;(2):CD003725. doi: 10.1002/14651858.CD003725.pub2. PMID 15106215
- [Background] Markham A, Bryson HM. Deflazacort. A review of its pharmacological properties and therapeutic efficacy. Drugs. 1995 Aug;50(2):317-33. doi: 10.2165/00003495-199550020-00008. PMID 8521761
- [Background] Markham LW, Spicer RL, Khoury PR, Wong BL, Mathews KD, Cripe LH. Steroid therapy and cardiac function in Duchenne muscular dystrophy. Pediatr Cardiol. 2005 Nov-Dec;26(6):768-71. doi: 10.1007/s00246-005-0909-4. PMID 15990951
- [Background] Mayhew A, Cano S, Scott E, Eagle M, Bushby K, Muntoni F; North Star Clinical Network for Paediatric Neuromuscular Disease. Moving towards meaningful measurement: Rasch analysis of the North Star Ambulatory Assessment in Duchenne muscular dystrophy. Dev Med Child Neurol. 2011 Jun;53(6):535-42. doi: 10.1111/j.1469-8749.2011.03939.x. Epub 2011 Mar 17. PMID 21410696
- [Background] Mendell JR, Moxley RT, Griggs RC, Brooke MH, Fenichel GM, Miller JP, King W, Signore L, Pandya S, Florence J, et al. Randomized, double-blind six-month trial of prednisone in Duchenne's muscular dystrophy. N Engl J Med. 1989 Jun 15;320(24):1592-7. doi: 10.1056/NEJM198906153202405. PMID 2657428
- [Background] Merlini L, Cicognani A, Malaspina E, Gennari M, Gnudi S, Talim B, Franzoni E. Early prednisone treatment in Duchenne muscular dystrophy. Muscle Nerve. 2003 Feb;27(2):222-7. doi: 10.1002/mus.10319. PMID 12548530
- [Background] Moxley RT 3rd, Ashwal S, Pandya S, Connolly A, Florence J, Mathews K, Baumbach L, McDonald C, Sussman M, Wade C; Quality Standards Subcommittee of the American Academy of Neurology; Practice Committee of the Child Neurology Society. Practice parameter: corticosteroid treatment of Duchenne dystrophy [RETIRED]: report of the Quality Standards Subcommittee of the American Academy of Neurology and the Practice Committee of the Child Neurology Society. Neurology. 2005 Jan 11;64(1):13-20. doi: 10.1212/01.WNL.0000148485.00049.B7. PMID 15642897
- [Background] O'Brien PC. Procedures for comparing samples with multiple endpoints. Biometrics. 1984 Dec;40(4):1079-87. PMID 6534410
- [Background] Phillips MF, Quinlivan RC, Edwards RH, Calverley PM. Changes in spirometry over time as a prognostic marker in patients with Duchenne muscular dystrophy. Am J Respir Crit Care Med. 2001 Dec 15;164(12):2191-4. doi: 10.1164/ajrccm.164.12.2103052. PMID 11751186
- [Background] Pocock SJ, Geller NL, Tsiatis AA. The analysis of multiple endpoints in clinical trials. Biometrics. 1987 Sep;43(3):487-98. PMID 3663814
- [Background] Quinlivan R, Roper H, Davie M, Shaw NJ, McDonagh J, Bushby K. Report of a Muscular Dystrophy Campaign funded workshop Birmingham, UK, January 16th 2004. Osteoporosis in Duchenne muscular dystrophy; its prevalence, treatment and prevention. Neuromuscul Disord. 2005 Jan;15(1):72-9. doi: 10.1016/j.nmd.2004.09.009. Epub 2004 Dec 10. No abstract available. PMID 15639124
- [Background] Reitter B. Deflazacort vs. prednisone in Duchenne muscular dystrophy: trends of an ongoing study. Brain Dev. 1995;17 Suppl:39-43. PMID 8882570
- [Background] Sansome A, Royston P, Dubowitz V. Steroids in Duchenne muscular dystrophy; pilot study of a new low-dosage schedule. Neuromuscul Disord. 1993 Sep-Nov;3(5-6):567-9. doi: 10.1016/0960-8966(93)90117-3. PMID 8186713
- [Background] Silversides CK, Webb GD, Harris VA, Biggar DW. Effects of deflazacort on left ventricular function in patients with Duchenne muscular dystrophy. Am J Cardiol. 2003 Mar 15;91(6):769-72. doi: 10.1016/s0002-9149(02)03429-x. No abstract available. PMID 12633823
- [Background] Simonds AK, Muntoni F, Heather S, Fielding S. Impact of nasal ventilation on survival in hypercapnic Duchenne muscular dystrophy. Thorax. 1998 Nov;53(11):949-52. doi: 10.1136/thx.53.11.949. PMID 10193393
- [Background] Stein RE, Jessop DJ. Functional status II(R). A measure of child health status. Med Care. 1990 Nov;28(11):1041-55. doi: 10.1097/00005650-199011000-00006. PMID 2250491
- [Background] Tang DI, Geller NL, Pocock SJ. On the design and analysis of randomized clinical trials with multiple endpoints. Biometrics. 1993 Mar;49(1):23-30. PMID 8513104
- [Background] Varni JW, Seid M, Knight TS, Uzark K, Szer IS. The PedsQL 4.0 Generic Core Scales: sensitivity, responsiveness, and impact on clinical decision-making. J Behav Med. 2002 Apr;25(2):175-93. doi: 10.1023/a:1014836921812. PMID 11977437
- [Background] Varni JW, Seid M, Kurtin PS. PedsQL 4.0: reliability and validity of the Pediatric Quality of Life Inventory version 4.0 generic core scales in healthy and patient populations. Med Care. 2001 Aug;39(8):800-12. doi: 10.1097/00005650-200108000-00006. PMID 11468499
- [Background] Varni JW, Seid M, Rode CA. The PedsQL: measurement model for the pediatric quality of life inventory. Med Care. 1999 Feb;37(2):126-39. doi: 10.1097/00005650-199902000-00003. PMID 10024117
- [Background] Witt WP, Kasper JD, Riley AW. Mental health services use among school-aged children with disabilities: the role of sociodemographics, functional limitations, family burdens, and care coordination. Health Serv Res. 2003 Dec;38(6 Pt 1):1441-66. doi: 10.1111/j.1475-6773.2003.00187.x. PMID 14727782
- [Background] Xie H, Heitjan DF. Sensitivity analysis of causal inference in a clinical trial subject to crossover. Clin Trials. 2004 Feb;1(1):21-30. doi: 10.1191/1740774504cn005oa. PMID 16281459
- [Derived] Guglieri M, Bushby K, McDermott MP, Hart KA, Tawil R, Martens WB, Herr BE, McColl E, Speed C, Wilkinson J, Kirschner J, King WM, Eagle M, Brown MW, Willis T, Griggs RC; FOR-DMD Investigators of the Muscle Study Group; Straub V, van Ruiten H, Childs AM, Ciafaloni E, Shieh PB, Spinty S, Maggi L, Baranello G, Butterfield RJ, Horrocks IA, Roper H, Alhaswani Z, Flanigan KM, Kuntz NL, Manzur A, Darras BT, Kang PB, Morrison L, Krzesniak-Swinarska M, Mah JK, Mongini TE, Ricci F, von der Hagen M, Finkel RS, O'Reardon K, Wicklund M, Kumar A, McDonald CM, Han JJ, Joyce N, Henricson EK, Schara-Schmidt U, Gangfuss A, Wilichowski E, Barohn RJ, Statland JM, Campbell C, Vita G, Vita GL, Howard JF Jr, Hughes I, McMillan HJ, Pegoraro E, Bello L, Burnette WB, Thangarajh M, Chang T. Effect of Different Corticosteroid Dosing Regimens on Clinical Outcomes in Boys With Duchenne Muscular Dystrophy: A Randomized Clinical Trial. JAMA. 2022 Apr 19;327(15):1456-1468. doi: 10.1001/jama.2022.4315. PMID 35381069
- [Derived] Schiava M, Amos R, VanRuiten H, McDermott MP, Martens WB, Gregory S, Mayhew A, McColl E, Tawil R, Willis T, Bushby K, Griggs RC, Guglieri M; FOR-DMD Investigators of the Muscle Study Group. Clinical and Genetic Characteristics in Young, Glucocorticoid-Naive Boys With Duchenne Muscular Dystrophy. Neurology. 2022 Jan 24;98(4):e390-e401. doi: 10.1212/WNL.0000000000013122. PMID 34857536

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 229 were screened for eligibility. 33 failed screening
Period: Overall Study
Arm/Group | Daily Prednisone | Daily Deflazacort | Intermittent Prednisone
Started | 65 | 65 | 66
Completed | 54 | 54 | 56
Not Completed | 11 | 11 | 10
Not completed — Adverse Event | 1 | 1 | 1
Not completed — Protocol Violation | 2 | 2 | 0
Not completed — Withdrawal by Subject | 8 | 5 | 7
Not completed — Lost to Follow-up | 0 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Daily Prednisone | Daily Deflazacort | Intermittent Prednisone | Total
Number analyzed (Participants) | 65 | 65 | 66 | 196
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.8 (1.0) | 5.8 (1.0) | 5.9 (1.1) | 5.9 (1.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 65 | 65 | 66 | 196
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 9 | 13 | 31
  Not Hispanic or Latino | 56 | 56 | 53 | 165
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 59 | 58 | 49 | 166
  race other than Caucasian | 6 | 7 | 17 | 30
Region of Enrollment [Number; unit: participants]
  Canada | 5 | 4 | 4 | 13
  United States | 27 | 27 | 28 | 82
  Italy | 8 | 7 | 7 | 22
  United Kingdom | 19 | 20 | 20 | 59
  Germany | 6 | 7 | 7 | 20
Mean weight [Mean (Standard Deviation); unit: kg] | 20.0 (3.0) | 19.9 (4.3) | 20.2 (3.5) | 20.0 (3.6)
Mean height [Mean (Standard Deviation); unit: cm] — Population: Data was not collected for one participant in the intermittent prednisone arm.
  cm
    number analyzed (Participants) | 65 | 65 | 65 | 195
    (all) | 109.9 (7.0) | 109.5 (7.6) | 110.9 (7.1) | 110.1 (7.2)
Mean body mass index [Mean (Standard Deviation); unit: kg/m^2] — Population: Data was not collected for one participant in the intermittent prednisone arm.
  kg/m^2
    number analyzed (Participants) | 65 | 65 | 65 | 195
    (all) | 16.5 (1.3) | 16.5 (2.0) | 16.4 (1.6) | 16.4 (1.6)
Mean rise from floor velocity [Mean (Standard Deviation); unit: rise/sec] | 0.19 (0.09) | 0.19 (0.07) | 0.18 (0.08) | 0.18 (0.08)
Mean 10 meter walk/run velocity [Mean (Standard Deviation); unit: 10 m/s] | 0.17 (0.04) | 0.17 (0.04) | 0.19 (0.04) | 0.17 (0.04)
Mean NSAA total score [Mean (Standard Deviation); unit: units on a scale] — The North Star Ambulatory Assessment (NSAA) is a 17-item rating scale that is used to measure functional motor abilities in ambulant children with Duchenne Muscular Dystrophy (DMD). It is usually used to monitor the progression of the disease and treatment effects.
  The activities are graded as follows:
  2 - "Normal" - no obvious modification of activity
  1 - Modified method but achieves goal independent of physical assistance from another 0 - Unable to achieve independently
  This scale is ordinal with 34 as the maximum score indicating fully-independent function.
  units on a scale | 22.0 (5.7) | 21.1 (5.7) | 21.1 (4.9) | 21.4 (5.4)
Mean Six-minute walk test distance [Mean (Standard Deviation); unit: meters] — Population: Data was not collected for two participants in the daily prednisone arm and one participant in the intermittent prednisone arm.
  meters
    number analyzed (Participants) | 63 | 65 | 65 | 193
    (all) | 342.4 (58.0) | 330.4 (65.1) | 331.6 (63.6) | 334.7 (62.2)
Mean forced vital capacity [Mean (Standard Deviation); unit: liters] | 1.0 (0.4) | 1.1 (0.4) | 1.1 (0.4) | 1.1 (0.4)
Mean percentage of predicted normal forced vital capacity [Mean (Standard Deviation); unit: percentage predicted normal] — Population: Data was not collected for one participant in the intermittent prednisone arm.
  percentage predicted normal
    number analyzed (Participants) | 65 | 65 | 65 | 195
    (all) | 85.4 (29.8) | 87.2 (36.2) | 88.1 (34.0) | 86.9 (33.3)

OUTCOME MEASURES:

1. Primary Outcome: Forced Vital Capacity
Description: Forced vital capacity was measured during a spirometry test. Forced expiratory volume (FEV) measures how much air a person can exhale during a forced breath. Forced vital capacity (FVC) is the total amount of air exhaled during the FEV test.
Time Frame: Average of Months 3, 6, 12, 18, 24, 30 and 36 visits
Population: Data was not collected on 4 participants in the daily prednisone arm, 3 participants in the deflazacort arm and 1 participant in the intermittent prednisone arm.
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Daily Prednisone | Daily Deflazacort | Intermittent Prednisone
Number analyzed (Participants) | 61 | 62 | 65
liters | 1.4 (0.03) | 1.4 (0.03) | 1.5 (0.03)
Statistical Analysis 1: Comparison: Daily Prednisone vs Daily Deflazacort; Test type: Superiority; p = 0.3904, Mixed Models Analysis
Statistical Analysis 2: Comparison: Daily Prednisone vs Intermittent Prednisone; Test type: Superiority; p = 0.5690, Mixed Models Analysis
Statistical Analysis 3: Comparison: Daily Prednisone vs Intermittent Prednisone; Test type: Superiority; p = 0.1518, Mixed Models Analysis

2. Primary Outcome: Rise From the Floor Velocity
Description: Reciprocal of time to rise from the floor
Time Frame: Average of Months 3, 6, 12, 18, 24, 30 and 36 visits
Population: Data was not collected on 3 participants in the daily prednisone arm, 2 participants in the deflazacort arm and 1 participant in the intermittent prednisone arm.
Measure: Least Squares Mean (Standard Error); unit: rise/sec
Arm/Group | Daily Prednisone | Daily Deflazacort | Intermittent Prednisone
Number analyzed (Participants) | 62 | 63 | 65
rise/sec | 0.24 (0.01) | 0.24 (0.01) | 0.18 (0.01)
Statistical Analysis 1: Comparison: Daily Prednisone vs Daily Deflazacort; Test type: Superiority; p = 0.7365, Mixed Models Analysis
Statistical Analysis 2: Comparison: Daily Prednisone vs Intermittent Prednisone; Test type: Superiority; p < 0.0001, Mixed Models Analysis
Statistical Analysis 3: Comparison: Daily Deflazacort vs Intermittent Prednisone; Test type: Superiority; p < 0.0001, Mixed Models Analysis

3. Primary Outcome: Treatment Satisfaction Questionnaire for Medication (TSQM) Global Satisfaction With Treatment Score
Description: The TSQM Global Satisfaction with Treatment is a 14-item questionnaire that ranges from 0 - 100 with higher scores indicating better outcomes.
Time Frame: Average of Months 3, 6, 12, 18, 24, 30 and 36 visits
Population: Data was not collected on 3 participants in the daily prednisone arm, 3 participants in the deflazacort arm and 1 participant in the intermittent prednisone arm.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Daily Prednisone | Daily Deflazacort | Intermittent Prednisone
Number analyzed (Participants) | 62 | 62 | 65
score on a scale | 71.2 (2.3) | 67.8 (2.3) | 65.1 (2.3)
Statistical Analysis 1: Comparison: Daily Prednisone vs Daily Deflazacort; Test type: Superiority; p = 0.2456, Mixed Models Analysis
Statistical Analysis 2: Comparison: Daily Prednisone vs Intermittent Prednisone; Test type: Superiority; p = 0.0369, Mixed Models Analysis
Statistical Analysis 3: Comparison: Daily Deflazacort vs Intermittent Prednisone; Test type: Superiority; p = 0.3589, Mixed Models Analysis

4. Secondary Outcome: North Star Ambulatory Assessment (NSAA) Score
Description: The North Star Ambulatory Assessment (NSAA) is a 17-item rating scale that is used to measure functional motor abilities in ambulant children with Duchenne Muscular Dystrophy (DMD). It is usually used to monitor the progression of the disease and treatment effects.
  The activities are graded as follows:
  2 - "Normal" - no obvious modification of activity
  1 - Modified method but achieves goal independent of physical assistance from another 0 - Unable to achieve independently This scale is ordinal with 34 as the maximum score indicating fully-independent function.
Time Frame: Average of Months 3, 6, 12, 18, 24, 30 and 36 visits
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Daily Prednisone | Daily Deflazacort | Intermittent Prednisone
Number analyzed (Participants) | 62 | 63 | 65
score on a scale | 23.7 (0.6) | 24.0 (0.6) | 20.7 (0.6)
Statistical Analysis 1: Comparison: Daily Prednisone vs Daily Deflazacort; Test type: Superiority; p = 0.7335, Mixed Models Analysis
Statistical Analysis 2: Comparison: Daily Prednisone vs Intermittent Prednisone; Test type: Superiority; p = 0.0004, Mixed Models Analysis
Statistical Analysis 3: Comparison: Daily Deflazacort vs Intermittent Prednisone; Test type: Superiority; p = 0.0001, Mixed Models Analysis

5. Secondary Outcome: 6 Minute Walk Test
Description: Measures the total distance walked in 6 minutes averaged over all post-baseline follow-up visits through Month 36.
Time Frame: Average of Months 3, 6, 12, 18, 24, 30 and 36 visits
Population: Data was not collected on 5 participants in the daily prednisone arm, 2 participants in the deflazacort arm and 2 participant in the intermittent prednisone arm.
Measure: Least Squares Mean (Standard Error); unit: meters
Arm/Group | Daily Prednisone | Daily Deflazacort | Intermittent Prednisone
Number analyzed (Participants) | 60 | 63 | 64
meters | 384.95 (9.6) | 384.17 (9.7) | 346.81 (9.4)
Statistical Analysis 1: Comparison: Daily Prednisone vs Daily Deflazacort; Test type: Superiority; p = 0.9532, Mixed Models Analysis
Statistical Analysis 2: Comparison: Daily Prednisone vs Intermittent Prednisone; Test type: Superiority; p = 0.0040, Mixed Models Analysis
Statistical Analysis 3: Comparison: Daily Deflazacort vs Intermittent Prednisone; Test type: Superiority; p = 0.0046, Mixed Models Analysis

6. Secondary Outcome: Range of Motion (Goniometry) of Left Ankle
Description: Range of motion at the ankle joint in dorsiflexion measured in degrees from plantigrade averaged over all post-baseline visits.
Time Frame: Average of Months 3, 6, 12, 18, 24, 30 and 36 visits
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Daily Prednisone | Daily Deflazacort | Intermittent Prednisone
Number analyzed (Participants) | 62 | 62 | 65
degrees | 4.39 (0.83) | 3.29 (0.85) | 2.67 (0.82)
Statistical Analysis 1: Comparison: Daily Prednisone vs Daily Deflazacort; Test type: Superiority; p = 0.3320, Mixed Models Analysis
Statistical Analysis 2: Comparison: Daily Prednisone vs Intermittent Prednisone; Test type: Superiority; p = 0.1248, Mixed Models Analysis
Statistical Analysis 3: Comparison: Daily Deflazacort vs Intermittent Prednisone; Test type: Superiority; p = 0.5854, Mixed Models Analysis

7. Secondary Outcome: Range of Motion (Goniometry) of Right Ankle
Description: as for outcome 6
Time Frame: Average of Months 3, 6, 12, 18, 24, 30 and 36 visits
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Daily Prednisone | Daily Deflazacort | Intermittent Prednisone
Number analyzed (Participants) | 62 | 62 | 65
degrees | 4.05 (0.89) | 2.81 (0.92) | 2.29 (0.89)
Statistical Analysis 1: Comparison: Daily Prednisone vs Daily Deflazacort; Test type: Superiority; p = 0.30814, Mixed Models Analysis
Statistical Analysis 2: Comparison: Daily Prednisone vs Intermittent Prednisone; Test type: Superiority; p = 0.1405, Mixed Models Analysis
Statistical Analysis 3: Comparison: Daily Deflazacort vs Intermittent Prednisone; Test type: Superiority; p = 0.6640, Mixed Models Analysis

8. Secondary Outcome: Number of Participants Who Tolerated the Regimen
Description: The number of participants who completed 36 months of follow-up on the originally assigned dosage (for weight) of study medication.
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Daily Prednisone | Daily Deflazacort | Intermittent Prednisone
Number analyzed (Participants) | 65 | 65 | 66
Participants | 36 | 36 | 37

9. Secondary Outcome: Heart Rate
Description: Measured by trans-thoracic echocardiogram and 12-lead ECG.
Time Frame: 36 months
Population: Data was not collected on 1 participant in the daily prednisone arm, and 2 participants in the intermittent prednisone arm.
Measure: Least Squares Mean (Standard Error); unit: bpm
Arm/Group | Daily Prednisone | Daily Deflazacort | Intermittent Prednisone
Number analyzed (Participants) | 64 | 65 | 64
bpm | 94.10 (1.96) | 93.52 (2.09) | 91.65 (2.10)
Statistical Analysis 1: Comparison: Daily Prednisone vs Daily Deflazacort; Test type: Superiority; p = 0.8345, Mixed Models Analysis
Statistical Analysis 2: Comparison: Daily Prednisone vs Intermittent Prednisone; Test type: Superiority; p = 0.3762, Mixed Models Analysis
Statistical Analysis 3: Comparison: Daily Deflazacort vs Intermittent Prednisone; Test type: Superiority; p = 0.5059, Mixed Models Analysis

10. Secondary Outcome: Quality of Life - Parent
Description: Quality of life was measured by parent/guardian self-report for all children utilizing the PEDSQL measurement tool. This is a 23-question tool. Scores can range from 0 to 100, with higher scores indicating better quality of life for the child.
Time Frame: Average of Months 12, 24, and 36 visits
Population: Data was not collected on 3 participants in the daily prednisone arm, 1 participants in the deflazacort arm and 2 participant in the intermittent prednisone arm.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Daily Prednisone | Daily Deflazacort | Intermittent Prednisone
Number analyzed (Participants) | 62 | 64 | 64
score on a scale | 64.88 (1.67) | 63.71 (1.69) | 61.33 (1.69)
Statistical Analysis 1: Comparison: Daily Prednisone vs Daily Deflazacort; Test type: Superiority; p = 0.5947, Mixed Models Analysis
Statistical Analysis 2: Comparison: Daily Prednisone vs Intermittent Prednisone; Test type: Superiority; p = 0.1098, Mixed Models Analysis
Statistical Analysis 3: Comparison: Daily Deflazacort vs Intermittent Prednisone; Test type: Superiority; p = 0.2803, Mixed Models Analysis

11. Secondary Outcome: Quality of Life- Child
Description: Quality of life was measured by child self-report in children age 5 and older utilizing the PEDSQL measurement tool. This is a 23-question tool. Scores can range from 0 to 100, with higher scores indicating better quality of life.
Time Frame: Average of Months 12, 24, and 36 visits
Population: Only children over the age of 5 self-reported quality of life.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Daily Prednisone | Daily Deflazacort | Intermittent Prednisone
Number analyzed (Participants) | 54 | 52 | 47
score on a scale | 67.39 (2.16) | 64.96 (2.17) | 65.07 (2.17)
Statistical Analysis 1: Comparison: Daily Prednisone vs Daily Deflazacort; Test type: Superiority; p = 0.3875, Mixed Models Analysis
Statistical Analysis 2: Comparison: Daily Prednisone vs Intermittent Prednisone; Test type: Superiority; p = 0.4240, Mixed Models Analysis
Statistical Analysis 3: Comparison: Daily Deflazacort vs Intermittent Prednisone; Test type: Superiority; p = 0.9683, Mixed Models Analysis

12. Secondary Outcome: Left Ventricular Ejection Fraction Percent
Description: Measured by trans-thoracic echocardiogram and 12-lead ECG.
Time Frame: 36 months
Population: Data was not collected on 2 participants in the daily prednisone arm, 3 participants in the deflazacort arm and 5 participants in the intermittent prednisone arm.
Measure: Least Squares Mean (Standard Error); unit: percentage of ejection fraction
Arm/Group | Daily Prednisone | Daily Deflazacort | Intermittent Prednisone
Number analyzed (Participants) | 63 | 62 | 61
percentage of ejection fraction | 61.88 (1.09) | 62.65 (1.17) | 62.45 (1.23)
Statistical Analysis 1: Comparison: Daily Prednisone vs Daily Deflazacort; Test type: Superiority; p = 0.6161, Mixed Models Analysis
Statistical Analysis 2: Comparison: Daily Prednisone vs Intermittent Prednisone; Test type: Superiority; p = 0.7302, Mixed Models Analysis
Statistical Analysis 3: Comparison: Daily Deflazacort vs Intermittent Prednisone; Test type: Superiority; p = 0.9007, Mixed Models Analysis

13. Secondary Outcome: Fractional Shortening Percent
Description: Measured by trans-thoracic echocardiogram and 12-lead ECG.
Time Frame: 36 months
Population: Data was not collected on 4 participants in the daily prednisone arm, 4 participants in the deflazacort arm and 8 participants in the intermittent prednisone arm.
Measure: Least Squares Mean (Standard Error); unit: percentage of fractional shortening
Arm/Group | Daily Prednisone | Daily Deflazacort | Intermittent Prednisone
Number analyzed (Participants) | 61 | 61 | 58
percentage of fractional shortening | 33.74 (0.81) | 34.01 (0.87) | 34.33 (0.87)
Statistical Analysis 1: Comparison: Daily Prednisone vs Daily Deflazacort; Test type: Superiority; p = 0.8138, Mixed Models Analysis
Statistical Analysis 2: Comparison: Daily Prednisone vs Intermittent Prednisone; Test type: Superiority; p = 0.5995, Mixed Models Analysis
Statistical Analysis 3: Comparison: Daily Deflazacort vs Intermittent Prednisone; Test type: Superiority; p = 0.7616, Mixed Models Analysis

14. Secondary Outcome: PR Interval
Description: Measured by trans-thoracic echocardiogram and 12-lead ECG.
Time Frame: 36 months
Population: Data was not collected on 3 participants in the daily prednisone arm, and 3 participants in the intermittent prednisone arm.
Measure: Least Squares Mean (Standard Error); unit: milliseconds
Arm/Group | Daily Prednisone | Daily Deflazacort | Intermittent Prednisone
Number analyzed (Participants) | 62 | 65 | 63
milliseconds | 115.59 (2.30) | 116.87 (2.33) | 117.90 (2.22)
Statistical Analysis 1: Comparison: Daily Prednisone vs Daily Deflazacort; Test type: Superiority; p = 0.6800, Mixed Models Analysis
Statistical Analysis 2: Comparison: Daily Prednisone vs Intermittent Prednisone; Test type: Superiority; p = 0.4365, Mixed Models Analysis
Statistical Analysis 3: Comparison: Daily Deflazacort vs Intermittent Prednisone; Test type: Superiority; p = 0.7281, Mixed Models Analysis

15. Secondary Outcome: Participant Weight
Time Frame: 36 months
Measure: Least Squares Mean (Standard Error); unit: kilograms
Arm/Group | Daily Prednisone | Daily Deflazacort | Intermittent Prednisone
Number analyzed (Participants) | 62 | 62 | 65
kilograms | 26.3 (0.36) | 24.9 (0.36) | 26.3 (0.35)
Statistical Analysis 1: Comparison: Daily Prednisone vs Daily Deflazacort; Test type: Superiority; p = 0.0041, Mixed Models Analysis; Mean Difference (Net) = -1.545, 98.3% CI 2-sided [-2.6611 to -0.2479]
Statistical Analysis 2: Comparison: Daily Prednisone vs Intermittent Prednisone; Test type: Superiority; p = 0.9076, Mixed Models Analysis; Mean Difference (Net) = 0.9076, 98.3% CI 2-sided [-1.248 to 1.1331]
Statistical Analysis 3: Comparison: Daily Deflazacort vs Intermittent Prednisone; Test type: Superiority; p = 0.0054, Mixed Models Analysis; Mean Difference (Net) = 1.3971, 98.3% CI 2-sided [0.2014 to 2.5927]

16. Secondary Outcome: Participant Height
Time Frame: 36 months
Measure: Least Squares Mean (Standard Error); unit: centimeters
Arm/Group | Daily Prednisone | Daily Deflazacort | Intermittent Prednisone
Number analyzed (Participants) | 62 | 62 | 65
centimeters | 116.8 (0.26) | 115.3 (0.27) | 119.9 (0.26)
Statistical Analysis 1: Comparison: Daily Prednisone vs Daily Deflazacort; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mean Difference (Net) = -1.48, 98.3% CI 2-sided [-2.3242 to -0.6358]
Statistical Analysis 2: Comparison: Daily Prednisone vs Intermittent Prednisone; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mean Difference (Net) = 3.054, 98.3% CI 2-sided [2.2222 to 3.8857]
Statistical Analysis 3: Comparison: Daily Deflazacort vs Intermittent Prednisone; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mean Difference (Net) = 4.534, 98.3% CI 2-sided [3.6941 to 5.3738]

17. Secondary Outcome: Participant Body Mass Index
Time Frame: 36 months
Measure: Least Squares Mean (Standard Error); unit: kilograms/square meter
Arm/Group | Daily Prednisone | Daily Deflazacort | Intermittent Prednisone
Number analyzed (Participants) | 62 | 62 | 65
kilograms/square meter | 18.9 (0.27) | 18.3 (0.26) | 18.1 (0.25)
Statistical Analysis 1: Comparison: Daily Prednisone vs Daily Deflazacort; Test type: Superiority; p = 0.0853, Mixed Models Analysis; Mean Difference (Net) = -0.6205, 98.3% CI 2-sided [-1.4845 to 0.2434]
Statistical Analysis 2: Comparison: Daily Prednisone vs Intermittent Prednisone; Test type: Superiority; p = 0.0143, Mixed Models Analysis; Mean Difference (Net) = -0.876, 98.3% CI 2-sided [-1.7292 to -0.0229]
Statistical Analysis 3: Comparison: Daily Deflazacort vs Intermittent Prednisone; Test type: Superiority; p = 0.4731, Mixed Models Analysis; Mean Difference (Net) = -0.2555, 98.3% CI 2-sided [-1.1117 to 0.6007]

ADVERSE EVENTS:
Time Frame: 36 months
Arm/Group | Daily Prednisone | Daily Deflazacort | Intermittent Prednisone
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/65 | 0/66
Serious Adverse Events (participants affected / at risk) | 5/65 | 10/65 | 5/66
Other Adverse Events (participants affected / at risk) | 61/65 | 58/65 | 55/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Daily Prednisone (N=65) | Daily Deflazacort (N=65) | Intermittent Prednisone (N=66)
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1
adenotonsillectomy (General disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Fetal Incontinence (Renal and urinary disorders) | 1 | 0 | 0
mildly increase urine calcium/creatinine ratio (Renal and urinary disorders) | 1 | 0 | 0
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
lower respiratory tract infection (Infections and infestations) | 1 | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Tentomy (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Appendicitis (Gastrointestinal disorders) | 0 | 1 | 0
Bone fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Chromaturia (Renal and urinary disorders) | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 1
Ear infection (Infections and infestations) | 0 | 1 | 0
Fall (General disorders) | 0 | 1 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 1 | 1
Joint pain (Metabolism and nutrition disorders) | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0
Myoglobinuria (Renal and urinary disorders) | 0 | 1 | 0
Tonsillitis (Blood and lymphatic system disorders) | 0 | 1 | 0
Oral Infection (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Circumsion (Reproductive system and breast disorders) | 0 | 0 | 1
Epistaxis (General disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Orchidopexy (Reproductive system and breast disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1
Umbilical hernia repair (Surgical and medical procedures) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Daily Prednisone (N=65) | Daily Deflazacort (N=65) | Intermittent Prednisone (N=66)
Cushingoid (Metabolism and nutrition disorders) | 6 | 6 | 3
Cataracts (Eye disorders) | 1 | 5 | 0
Vomiting (Gastrointestinal disorders) | 19 | 16 | 15
Diarrhea (Gastrointestinal disorders) | 9 | 7 | 10
Abdominal pain (Gastrointestinal disorders) | 8 | 8 | 8
Abdominal pain upper (Gastrointestinal disorders) | 10 | 4 | 10
Constipation (Gastrointestinal disorders) | 7 | 9 | 7
Nausea (Gastrointestinal disorders) | 5 | 4 | 1
Gastroenteritis (Gastrointestinal disorders) | 4 | 3 | 1
Abdominal discomfort (Gastrointestinal disorders) | 4 | 1 | 2
Gastrointestinal disorders (Gastrointestinal disorders) | 4 | 2 | 0
Pyrexia (General disorders) | 12 | 11 | 10
Malaise (General disorders) | 2 | 4 | 2
Ear infection (Infections and infestations) | 4 | 7 | 8
Influenza (Infections and infestations) | 8 | 1 | 2
Nasopharyngitis (Infections and infestations) | 4 | 2 | 2
Fall (Injury, poisoning and procedural complications) | 10 | 7 | 12
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 4 | 1
Abnormal weight gain (Metabolism and nutrition disorders) | 9 | 4 | 5
Vitamin D deficiency (Metabolism and nutrition disorders) | 7 | 6 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 10 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 6 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 6 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 5 | 3
Intervertebral disc space narrowing (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 1 | 0
Headache (Nervous system disorders) | 9 | 9 | 6
Abnormal behavior (Psychiatric disorders) | 12 | 17 | 16
Mood altered (Psychiatric disorders) | 4 | 7 | 2
Aggression (Psychiatric disorders) | 4 | 4 | 2
Insomnia (Psychiatric disorders) | 1 | 4 | 2
Psychomotor hyperactivity (Psychiatric disorders) | 2 | 1 | 4
Pollakiuria (Renal and urinary disorders) | 4 | 2 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 12 | 11
Naspharyngitis (Respiratory, thoracic and mediastinal disorders) | 9 | 9 | 11
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 11 | 11 | 7
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 6
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 2
Hypertrichosis (Skin and subcutaneous tissue disorders) | 5 | 7 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI cannot publish any manuscript without review and written consent of the FOR-DMD study steering committee.

DOCUMENTS (2):
  • Study Protocol (2019-12-18): https://cdn.clinicaltrials.gov/large-docs/07/NCT01603407/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-16): https://cdn.clinicaltrials.gov/large-docs/07/NCT01603407/SAP_001.pdf